CLINICAL TRIAL: NCT03999996
Title: A Phase 3, Follow-Up Trial to Evaluate Long-Term Safety and Antibody Persistence, and the Impact of a Booster Dose of a Tetravalent Dengue Vaccine Candidate in Healthy Adolescents and Adults in Areas Non-Endemic for Dengue
Brief Title: Long-Term Safety and Antibody Persistence of TDV and the Impact of a Booster Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEN-303; 2023-000027-36 (EudraCT Number)
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Dengue Fever
Keywords: Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded, randomized, and placebo-controlled from Month 15 onwards for participants from parent trial DEN-304 (US) and from Month 42 onwards for participants from parent trial DEN-315 (Mexico).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Prior to Booster: DEN-304 (Experimental): Participants who received TDV in parent trial DEN-304 (US) were assessed before they received booster dose (Placebo/TDV) at Month 15.
  Interventions: Biological: Takeda's Dengue Tetravalent Vaccine (Live, Attenuated) (TDV)
- Prior to Booster: DEN-315 (Experimental): Participants who received TDV in parent trial DEN-315 (Mexico) were assessed before they received booster dose (Placebo/TDV) at Month 42.
  Interventions: Biological: Takeda's Dengue Tetravalent Vaccine (Live, Attenuated) (TDV)
- Booster Phase: Placebo (Placebo Comparator): Participants received TDV placebo-matching 0.5 milliliters (ml) injection, subcutaneous (SC), once at Month 15 for participants from parent trial DEN-304 (US) or once at Month 42 for participants from parent trial DEN-315 (Mexico).
  Interventions: Biological: Placebo
- Booster Phase: TDV (Experimental): Participants received TDV 0.5 ml, injection, SC, once at Month 15 for participants from parent trial DEN-304 (US) or once at Month 42 for participants from parent trial DEN-315 (Mexico).
  Interventions: Biological: Takeda's Dengue Tetravalent Vaccine (Live, Attenuated) (TDV)

INTERVENTIONS:
Biological: Takeda's Dengue Tetravalent Vaccine (Live, Attenuated) (TDV) — TDV subcutaneous injection
  Arms: Booster Phase: TDV; Prior to Booster: DEN-304; Prior to Booster: DEN-315
Biological: Placebo — Normal Saline (0.9% NaCl) subcutaneous injection
  Arms: Booster Phase: Placebo

SUMMARY:
The purpose of this study is to describe antibody persistence for each of the 4 dengue serotypes for up to 63 months after the first vaccination in the primary vaccination series for participants from parent trial DEN-315 (NCT03341637) (Mexico) and for up to 36 months after the first vaccination in the primary vaccination series for participants from parent trial DEN-304 (NCT03423173) (United States [US]) and to describe the impact of a tetravalent dengue vaccine (TDV) booster dose vs placebo on antibody response for each of the 4 dengue serotypes at 1 month and 6 months post administration of the TDV booster or placebo.

DETAILED DESCRIPTION:
The vaccine tested in this study is Takeda's Dengue Tetravalent Vaccine (Live, Attenuated) (TDV). This study will look at the long-term antibody persistence and safety of Takeda's TDV in healthy adolescents and adults and will assess the impact of a booster dose.

The study has enrolled 365 healthy participants. Participants who previously received TDV in two parent trials (DEN-304 [NCT03423173] and DEN-315 [NCT03341637]), will be invited to participate in this follow-up trial. Participants will be assessed for antibody persistence and safety from Baseline (Month 0) through Month 15 (for participants from parent trial DEN-304 [US]) or Month 42 (for participants from parent trial DEN-315 [Mexico]). At Month 15 (for participants from parent trial DEN-304 [US]) or at Month 42 (for participants from parent trial DEN-315 [Mexico]), eligible participants will be randomized in 1:1 ratio to one of two trial groups to receive TDV or placebo:

A. Group 1- TDV 0.5 mL subcutaneous (SC) injection at Month 15 for participants from parent trial DEN-304 (US) or at Month 42 for participants from parent trial DEN-315 (Mexico]).

B. Group 2- Takeda's tetravalent dengue placebo (dummy SC injection - this is a liquid that looks like the study drug but has no active ingredient), 0.5 mL, subcutaneous injection at Month 15 for participants from parent trial DEN-304 (US) or at Month 42 for participants from parent trial DEN-315 (Mexico).

This multi-centre trial will be conducted in US and Mexico. The overall time to participate in this study is up to 21 months for parent trial DEN-304 (US) and up to 48 months for parent trial DEN-315 (Mexico). Participants from parent trial DEN-304 (US) and participants from parent trial DEN-315 (Mexico) will come for 5 visits to the clinic which includes a final visit (Visit 5) 6 months after the booster dose for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants (irrespective of serostatus at baseline in the parent trials (DEN-304 [(NCT03423173)] and DEN-315 [NCT03341637]) who received at least one dose of Takeda's tetravalent dengue vaccine candidate (TDV) in the parent trials and have data from at least one blood draw post-vaccination.

Exclusion Criteria:

1. Participants with a prolonged period of habitation (≥1 year) in a dengue endemic area within the 2 years prior to Visit 1 Day 1 (Month 0).
2. Previous and planned vaccination (during the trial conduct), against any flavivirus including dengue (other than Takeda's TDV), yellow fever (YF), Japanese encephalitis (JE) viruses or tick-borne encephalitis.

Booster Exclusion Criteria:

1. Participants for whom baseline serostatus is not defined in the parent trials (DEN-304 [(NCT03423173)] and DEN-315 [NCT03341637]).
2. Participants with any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (eg, Guillain-Barré syndrome).
3. Known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Month 42 for participants from parent trial DEN-315 (Mexico)/ Month 15 for participants from parent trial DEN-304 (US); use of inhaled, intranasal, or topical corticosteroids is allowed.
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Month 42 for participants from parent trial DEN-315 (Mexico)/ Month 15 for participants from parent trial DEN-304 (US).
   3. Administration of immunoglobulins and/or any blood products within the 3 months prior to administration of the TDV booster or placebo at Month 42 for participants from parent trial DEN-315 (Mexico)/ Month 15 for participants from parent trial DEN-304 (US); consider whether applicable as an exclusion criterion or criterion for delay.
   4. Receipt of immunostimulants within 60 days prior to Month 42 for participants from parent trial DEN-315 (Mexico)/ Month 15 for participants from parent trial DEN-304 (US).
   5. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Month 42 for participants from parent trial DEN-315 (Mexico) / Month 15 for participants from parent trial DEN-304 (US).
   6. Known human immunodeficiency virus (HIV) infection or HIV-related disease.
   7. Hepatitis C virus infection.
   8. Genetic immunodeficiency.
4. Abnormalities of splenic or thymic function.
5. Participants with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
6. Participants with history of current or previous infection with a flavivirus such as dengue, Zika, YF, JE, West Nile fever, tick-borne encephalitis or Murray Valley encephalitis and participants with a prolonged period of habitation (≥1 year) in a dengue endemic area during trial conduct.

Ages: 13 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 365 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (10):
- United States (8):
  - AES - DRS - Optimal Research Alabama - Huntsville, Huntsville, Alabama
  - AES - DRS - Optimal Research Illinois - Peoria, Peoria, Illinois
  - Alliance for Multispecialty Research, LLC - Newton - PPDS, Newton, Kansas
  - Optima Research, Rockville, Maryland
  - AES - DRS - Synexus Clinical Research US, Inc. Minneapolis, Richfield, Minnesota
  - AES - DRS - Synexus Clinical Research US, Inc. - St. Louis, St Louis, Missouri
  - AES - DRS - Synexus Clinical Research US, Inc. - Omaha, Papillion, Nebraska
  - Advanced Clinical Research/Velocity Clinical Research, West Jordan, Utah
- Mexico (2):
  - Instituto Nacional de Pediatria, Mexico City
  - CAIMED Investigacion en Salud S.A de C.V., Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a33e?idFilter=%5B%22DEN-303%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at multiple investigative sites in United States (US) and Mexico from 12 November 2019 to 25 May 2024.
Pre-assignment Details: Healthy participants who received Takeda's Dengue Tetravalent Vaccine (TDV) in two parent trials, DEN-304 [NCT03423173] and DEN-315 [NCT03341637] were enrolled to receive either placebo or TDV.
Groups:
- Prior to Booster: DEN-304: Participants who received TDV in parent trial DEN-304 (US) were assessed before they received booster dose (Placebo/TDV) at Visit 3 (Month 15).
- Prior to Booster: DEN-315: Participants who received TDV in parent trial DEN-315 (Mexico) were assessed before they received booster dose (Placebo/TDV) at Visit 3 (Month 42).
- Booster Phase: Placebo: Participants received TDV placebo-matching 0.5 milliliters (ml) injection, subcutaneous (SC), once at Visit 3 (Month 15) for participants from parent trial DEN-304 (US) or once at Visit 3 (Month 42) for participants from parent trial DEN-315 (Mexico).
- Booster Phase: TDV: Participants received TDV 0.5 ml, injection, SC, once at Visit 3 (Month 15) for participants from parent trial DEN-304 (US) or once at Visit 3 (Month 42) for participants from parent trial DEN-315 (Mexico).
Period: Prior to Booster
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315 | Booster Phase: Placebo | Booster Phase: TDV
Started | 246 | 119 | 0 | 0
Completed | 149 | 84 | 0 | 0
Not Completed | 97 | 35 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 22 | 0 | 0
Not completed — Withdrawal of Consent | 51 | 8 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Reason Not Specified | 27 | 4 | 0 | 0
Period: Booster Phase
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315 | Booster Phase: Placebo | Booster Phase: TDV
Started | 0 | 0 | 118 | 115
Completed | 0 | 0 | 115 | 110
Not Completed | 0 | 0 | 3 | 5
Not completed — Lost to Follow-up | 0 | 0 | 3 | 3
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 1
Not completed — Reason Not Specified | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set (SAF) included all participants who agreed to participate in the current trial, did not screen fail, and who received at least one dose of Takeda's TDV in the parent trials.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315 | Total
Number analyzed (Participants) | 246 | 119 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.03) | 16.3 (1.77) | 35.2 (16.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 70 | 215
  Male | 101 | 49 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 119 | 127
  Not Hispanic or Latino | 238 | 0 | 238
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 35 | 0 | 35
  White | 201 | 0 | 201
  More than one race | 4 | 117 | 121
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 1 (Month 0 [Day 1])
Description: GMTs of neutralizing antibodies were measured by microneutralization test 50% (MNT50) for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 1 at Month 0 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 0 (Day 1)
Population: Per Protocol Set (PPS) included all participants from the Full Analysis Set (FAS) who received two doses of Takeda's TDV in the parent trials with no new major protocol violations in this trial prior to administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
titer
  DENV-1 | 76.8 [62.0 to 95.2] | 88.6 [70.4 to 111.5]
  DENV-2 | 539.6 [460.9 to 631.7] | 425.6 [352.7 to 513.5]
  DENV-3 | 33.7 [28.0 to 40.5] | 29.5 [24.1 to 36.1]
  DENV-4 | 40.0 [33.1 to 48.4] | 27.1 [21.9 to 33.6]

2. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 2 (Month 12)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 2 at Month 12 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 12
Population: PPS included all participants from the FAS who received two doses of Takeda's TDV in the parent trials with no new major protocol violations in this trial prior to administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial. Overall number of participants analyzed: number of participants with data available for analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 182 | 48
titer
  DENV-1 | 58.4 [45.0 to 75.7] | 96.4 [69.9 to 132.7]
  DENV-2 | 427.3 [360.2 to 507.0] | 276.1 [208.3 to 365.9]
  DENV-3 | 32.8 [26.5 to 40.4] | 25.3 [18.5 to 34.7]
  DENV-4 | 30.0 [24.4 to 37.0] | 22.9 [17.6 to 29.8]

3. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 3 (Month 15) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 3 at Month 15 for participants from parent trial DEN-304.
Time Frame: Month 15 (DEN-304)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-304
Number analyzed (Participants) | 171
titer
  DENV-1 | 121.7 [93.3 to 158.7]
  DENV-2 | 560.2 [473.9 to 662.2]
  DENV-3 | 40.3 [32.6 to 49.8]
  DENV-4 | 34.1 [27.3 to 42.6]

4. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 3 (Month 42) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 3 at Month 42 for participants from parent trial DEN-315.
Time Frame: Month 42 (DEN-315)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-315
Number analyzed (Participants) | 80
titer
  DENV-1 | 106.5 [80.8 to 140.4]
  DENV-2 | 202.9 [159.5 to 258.2]
  DENV-3 | 21.9 [16.8 to 28.5]
  DENV-4 | 11.2 [9.1 to 13.6]

5. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 1 (Month 0 [Day 1])
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 1 at Month 0 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 0 [Day 1)
Population: PPS included all participants from the FAS who received two doses of Takeda's TDV in the parent trials with no new major protocol violations in this trial prior to administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial. Number analyzed: number of participants with data available for analysis for the specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
titer
  Parent Trial Baseline Serostatus:Positive: DENV-1: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive: DENV-1 | 122.8 [59.5 to 253.2] | 259.3 [135.7 to 495.5]
  Parent Trial Baseline Serostatus:Positive: DENV-2: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive: DENV-2 | 560.1 [314.3 to 998.1] | 714.1 [355.2 to 1435.7]
  Parent Trial Baseline Serostatus:Positive: DENV-3: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive: DENV-3 | 48.2 [26.1 to 88.9] | 118.7 [28.3 to 497.3]
  Parent Trial Baseline Serostatus:Positive: DENV-4: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive: DENV-4 | 61.5 [32.1 to 118.2] | 112.4 [29.6 to 427.5]
  Parent Trial Baseline Serostatus:Negative; DENV-1: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-1 | 71.3 [57.2 to 88.9] | 82.0 [64.7 to 103.9]
  Parent Trial Baseline Serostatus:Negative; DENV-2: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-2 | 536.4 [456.9 to 629.6] | 410.0 [337.1 to 498.6]
  Parent Trial Baseline Serostatus:Negative; DENV-3: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-3 | 31.8 [26.3 to 38.5] | 26.7 [22.1 to 32.2]
  Parent Trial Baseline Serostatus:Negative; DENV-4: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-4 | 37.3 [30.7 to 45.4] | 24.5 [19.9 to 30.0]

6. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 2 (Month 12)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 2 at Month 12 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 12
Population: PPS included all participants from the FAS who received two doses of Takeda's TDV in the parent trials with no new major protocol violations in this trial prior to administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial. Overall number of participants analyzed: number of participants with data available for analyses. Number analyzed: number of participants with data available for analysis for the specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 182 | 48
titer
  Parent Trial Baseline Serostatus:Positive; DENV-1: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-1 | 87.2 [37.2 to 204.4] | 93.5 [0.0 to 6220000]
  Parent Trial Baseline Serostatus:Positive; DENV-2: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-2 | 544.5 [279.1 to 1062.4] | 272.6 [0.0 to 12600000]
  Parent Trial Baseline Serostatus:Positive; DENV-3: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-3 | 48.6 [23.2 to 101.6] | 34.0 [9.99 to 99.9]
  Parent Trial Baseline Serostatus:Positive; DENV-4: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-4 | 48.0 [22.2 to 104.0] | 21.5 [16.0 to 28.9]
  Parent Trial Baseline Serostatus:Negative; DENV-1: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-1 | 54.8 [41.7 to 71.9] | 96.5 [69.3 to 134.2]
  Parent Trial Baseline Serostatus:Negative; DENV-2: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-2 | 411.1 [346.6 to 487.6] | 276.2 [206.7 to 369.0]
  Parent Trial Baseline Serostatus:Negative; DENV-3: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-3 | 30.8 [24.8 to 38.2] | 25.0 [18.0 to 34.7]
  Parent Trial Baseline Serostatus:Negative; DENV-4: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-4 | 27.8 [22.6 to 34.4] | 23.0 [17.5 to 30.2]

7. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 15) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 3 at Month 15 for participants from parent trial DEN-304.
Time Frame: Month 15 (DEN-304)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-304
Number analyzed (Participants) | 171
titer
  Parent Trial Baseline Serostatus:Positive; DENV-1: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive; DENV-1 | 214.3 [80.6 to 569.9]
  Parent Trial Baseline Serostatus:Positive; DENV-2: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive; DENV-2 | 484.5 [263.4 to 891.3]
  Parent Trial Baseline Serostatus:Positive; DENV-3: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive; DENV-3 | 60.4 [29.9 to 122.1]
  Parent Trial Baseline Serostatus:Positive; DENV-4: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive; DENV-4 | 47.0 [21.7 to 102.1]
  Parent Trial Baseline Serostatus:Negative; DENV-1: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative; DENV-1 | 110.9 [84.9 to 145.0]
  Parent Trial Baseline Serostatus:Negative; DENV-2: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative; DENV-2 | 573.6 [483.5 to 680.4]
  Parent Trial Baseline Serostatus:Negative; DENV-3: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative; DENV-3 | 37.7 [30.3 to 46.9]
  Parent Trial Baseline Serostatus:Negative; DENV-4: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative; DENV-4 | 32.4 [25.7 to 40.7]

8. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 42) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 3 at Month 42 for participants from parent trial DEN-315.
Time Frame: Month 42 (DEN-315)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Prior to Booster: DEN-315
Number analyzed (Participants) | 80
titer
  Parent Trial Baseline Serostatus:Positive; DENV-1: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive; DENV-1 | 320.0 [119.6 to 856.4]
  Parent Trial Baseline Serostatus:Positive; DENV-2: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive; DENV-2 | 436.6 [156.3 to 1219.1]
  Parent Trial Baseline Serostatus:Positive; DENV-3: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive; DENV-3 | 80.4 [17.5 to 369.3]
  Parent Trial Baseline Serostatus:Positive; DENV-4: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive; DENV-4 | 23.3 [4.3 to 125.1]
  Parent Trial Baseline Serostatus:Negative; DENV-1: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus:Negative; DENV-1 | 95.8 [72.2 to 127.2]
  Parent Trial Baseline Serostatus:Negative; DENV-2: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus:Negative; DENV-2 | 188.6 [147.3 to 241.4]
  Parent Trial Baseline Serostatus:Negative; DENV-3: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus:Negative; DENV-3 | 19.3 [15.1 to 24.8]
  Parent Trial Baseline Serostatus:Negative; DENV-4: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus:Negative; DENV-4 | 10.4 [8.8 to 12.4]

9. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 1 (Month 0 [Day 1])
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 1 at Month 0 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 0 (Day 1)
Population: PPS included all participants from the FAS who received two doses of Takeda's TDV in the parent trials with no new major protocol violations in this trial prior to administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
percentage of participants
  DENV-1 | 85.8 [80.7 to 89.9] | 92.4 [86.1 to 96.5]
  DENV-2 | 98.7 [96.4 to 99.7] | 99.2 [95.4 to 100]
  DENV-3 | 72.4 [66.3 to 78.0] | 79.8 [71.5 to 86.6]
  DENV-4 | 80.8 [75.2 to 85.6] | 76.5 [67.8 to 83.8]

10. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 2 (Month 12)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 2 at Month 12 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 182 | 48
percentage of participants
  DENV-1 | 78.6 [71.9 to 84.3] | 97.9 [88.9 to 100]
  DENV-2 | 100 [98.0 to 100] | 100 [92.6 to 100]
  DENV-3 | 72.0 [64.9 to 78.4] | 75.0 [60.4 to 86.4]
  DENV-4 | 76.4 [69.5 to 82.3] | 83.3 [69.8 to 92.5]

11. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity Rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 15 for participants from parent trial DEN-304.
Time Frame: Month 15 (DEN-304)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304
Number analyzed (Participants) | 171
percentage of participants
  DENV-1 | 94.2 [89.5 to 97.2]
  DENV-2 | 99.4 [96.8 to 100]
  DENV-3 | 81.9 [75.3 to 87.3]
  DENV-4 | 76.0 [68.9 to 82.2]

12. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster at Visit 3 (Month 42) (DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 42 for parent trial DEN-315.
Time Frame: Month 42 (DEN-315)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-315
Number analyzed (Participants) | 80
percentage of participants
  DENV-1 | 96.3 [89.4 to 99.2]
  DENV-2 | 98.8 [93.2 to 100]
  DENV-3 | 71.3 [60.0 to 80.8]
  DENV-4 | 55.0 [43.5 to 66.2]

13. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 1 [Month 0 (Day 1])
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 1 at Month 0 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 0 (Day 1)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
percentage of participants
  Parent Trial Baseline Serostatus:Positive; DENV-1: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive; DENV-1 | 81.8 [64.5 to 93.0] | 100 [63.1 to 100]
  Parent Trial Baseline Serostatus:Positive; DENV-2: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive; DENV-2 | 97.0 [84.2 to 100] | 100 [63.1 to 100]
  Parent Trial Baseline Serostatus:Positive; DENV-3: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive; DENV-3 | 75.8 [57.7 to 88.9] | 100 [63.1 to 100]
  Parent Trial Baseline Serostatus:Positive; DENV-4: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus:Positive; DENV-4 | 87.9 [71.8 to 96.6] | 100 [63.1 to 100]
  Parent Trial Baseline Serostatus:Negative; DENV-1: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-1 | 86.4 [81.0 to 90.8] | 91.9 [85.2 to 96.2]
  Parent Trial Baseline Serostatus:Negative; DENV-2: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-2 | 99.0 [96.5 to 99.9] | 99.1 [95.1 to 100]
  Parent Trial Baseline Serostatus:Negative; DENV-3: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-3 | 71.8 [65.2 to 77.9] | 78.4 [69.6 to 85.6]
  Parent Trial Baseline Serostatus:Negative; DENV-4: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus:Negative; DENV-4 | 79.6 [73.5 to 84.9] | 74.8 [65.6 to 82.5]

14. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 2 (Month 12)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 2 at Month 12 for participants from both parent trials (DEN-304 and DEN-315).
Time Frame: Month 12
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 182 | 48
percentage of participants
  Parent Trial Baseline Serostatus:Positive; DENV-1: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-1 | 80.0 [59.3 to 93.2] | 100 [15.8 to 100]
  Parent Trial Baseline Serostatus:Positive; DENV-2: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-2 | 100 [86.3 to 100] | 100 [15.8 to 100]
  Parent Trial Baseline Serostatus:Positive; DENV-3: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-3 | 76.0 [54.9 to 90.6] | 100 [15.8 to 100]
  Parent Trial Baseline Serostatus:Positive; DENV-4: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus:Positive; DENV-4 | 80.0 [59.3 to 93.2] | 100 [15.8 to 100]
  Parent Trial Baseline Serostatus:Negative; DENV-1: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-1 | 78.3 [71.1 to 84.5] | 97.8 [88.5 to 100]
  Parent Trial Baseline Serostatus:Negative; DENV-2: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-2 | 100 [97.7 to 100] | 100 [92.3 to 100]
  Parent Trial Baseline Serostatus:Negative; DENV-3: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-3 | 71.3 [63.6 to 78.3] | 73.9 [58.9 to 85.7]
  Parent Trial Baseline Serostatus:Negative; DENV-4: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus:Negative; DENV-4 | 75.8 [68.3 to 82.3] | 82.6 [68.6 to 92.2]

15. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 15 for participants from parent trial DEN-304.
Time Frame: Month 15 (DEN-304)
Population: PPS included all participants from the FAS who received two doses of Takeda's TDV in the parent trials with no new major protocol violations in this trial prior to administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial Overall number of participants analyzed: number of participants with data available for analyses. Number analyzed: number of participants with data available for analysis for the specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304
Number analyzed (Participants) | 171
percentage of participants
  Parent Trial Baseline Serostatus:Positive; DENV-1: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive; DENV-1 | 87.5 [67.6 to 97.3]
  Parent Trial Baseline Serostatus:Positive; DENV-2: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive; DENV-2 | 100 [85.8 to 100]
  Parent Trial Baseline Serostatus:Positive; DENV-3: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive; DENV-3 | 83.3 [62.6 to 95.3]
  Parent Trial Baseline Serostatus:Positive: DENV-4: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus:Positive: DENV-4 | 79.2 [57.8 to 92.9]
  Parent Trial Baseline Serostatus:Negative: DENV-1: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative: DENV-1 | 95.2 [90.4 to 98.1]
  Parent Trial Baseline Serostatus:Negative: DENV-2: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative: DENV-2 | 99.3 [96.3 to 100]
  Parent Trial Baseline Serostatus:Negative: DENV-3: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative: DENV-3 | 81.6 [74.4 to 87.5]
  Parent Trial Baseline Serostatus:Negative: DENV-4: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus:Negative: DENV-4 | 75.5 [67.7 to 82.2]

16. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 42) ((DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 42 for parent trial DEN-315.
Time Frame: Month 42 (DEN-315)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-315
Number analyzed (Participants) | 80
percentage of participants
  Parent Trial Baseline Serostatus:Positive: DENV-1: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive: DENV-1 | 100 [59.0 to 100]
  Parent Trial Baseline Serostatus:Positive: DENV-2: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive: DENV-2 | 100 [59.0 to 100]
  Parent Trial Baseline Serostatus:Positive: DENV-3: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive: DENV-3 | 100 [59.0 to 100]
  Parent Trial Baseline Serostatus:Positive: DENV-4: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus:Positive: DENV-4 | 57.1 [18.4 to 90.1]
  Parent Trial Baseline Serostatus:Negative: DENV-1: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus:Negative: DENV-1 | 95.9 [88.5 to 99.1]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 98.6 [92.6 to 100]
  Parent Trial Baseline Serostatus; Negative:DENV-3: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus; Negative:DENV-3 | 68.5 [56.6 to 78.9]
  Parent Trial Baseline Serostatus; Negative: DENV-4: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus; Negative: DENV-4 | 54.8 [42.7 to 66.5]

17. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster at Visit 1 (Month 0 [Day 1])
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 1 at Month 0 for both parent trials (DEN-304 and DEN-315).
Time Frame: Month 0 (Day 1)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
percentage of participants
  Bivalent | 10.9 [7.2 to 15.5] | 9.2 [4.7 to 15.9]
  Trivalent | 20.5 [15.6 to 26.2] | 18.5 [12.0 to 26.6]
  Tetravalent | 61.9 [55.4 to 68.1] | 67.2 [58.0 to 75.6]

18. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster at Visit 2 (Month 12)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 2 at Month 12 for both parent trials (DEN-304 and DEN-315).
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 182 | 48
percentage of participants
  Bivalent | 12.6 [8.2 to 18.4] | 10.4 [3.5 to 22.7]
  Trivalent | 21.4 [15.7 to 28.1] | 22.9 [12.0 to 37.3]
  Tetravalent | 57.1 [49.6 to 64.4] | 66.7 [51.6 to 79.6]

19. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 15 for parent trial DEN-304.
Time Frame: Month 15 (DEN-304)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304
Number analyzed (Participants) | 171
percentage of participants
  Bivalent | 10.5 [6.4 to 16.1]
  Trivalent | 17.0 [11.7 to 23.4]
  Tetravalent | 69.0 [61.5 to 75.8]

20. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster at Visit 3 (Month 42) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 42 for parent trial DEN-315.
Time Frame: Month 42 (DEN-315)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-315
Number analyzed (Participants) | 80
percentage of participants
  Bivalent | 20.0 [11.9 to 30.4]
  Trivalent | 27.5 [18.1 to 38.6]
  Tetravalent | 48.8 [37.4 to 60.2]

21. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 1 (Month 0 [Day 1])
Description: as for outcome 17
Time Frame: Month 0 (Day 1)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
percentage of participants
  Parent Trial Baseline Serostatus;Positive: Bivalent: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus;Positive: Bivalent | 9.1 [1.9 to 24.3] | 0 [0.0 to 36.9]
  Parent Trial Baseline Serostatus;Positive: Trivalent: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus;Positive: Trivalent | 12.1 [3.4 to 28.2] | 0 [0.0 to 36.9]
  Parent Trial Baseline Serostatus;Positive: Tetravalent: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus;Positive: Tetravalent | 69.7 [51.3 to 84.4] | 100 [63.1 to 100]
  Parent Trial Baseline Serostatus;Negative: Bivalent: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus;Negative: Bivalent | 11.2 [7.2 to 16.3] | 9.9 [5.1 to 17.0]
  Parent Trial Baseline Serostatus;Negative: Trivalent: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus;Negative: Trivalent | 21.8 [16.4 to 28.1] | 19.8 [12.9 to 28.5]
  Parent Trial Baseline Serostatus;Negative: Tetravalent: number analyzed (Participants) | 206 | 111
  Parent Trial Baseline Serostatus;Negative: Tetravalent | 60.7 [53.7 to 67.4] | 64.9 [55.2 to 73.7]

22. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 2 (Month 12)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 2 at Month 12 for both parent trials (DEN-304 and DEN-315).
Time Frame: Month 12
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 182 | 48
percentage of participants
  Parent Trial Baseline Serostatus;Positive:Bivalent: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus;Positive:Bivalent | 4.0 [0.1 to 20.4] | 0 [0.0 to 84.2]
  Parent Trial Baseline Serostatus;Positive:Trivalent: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus;Positive:Trivalent | 20.0 [6.8 to 40.7] | 0 [0.0 to 84.2]
  Parent Trial Baseline Serostatus;Positive:Tetravalent: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus;Positive:Tetravalent | 64.0 [42.5 to 82.0] | 100 [15.8 to 100]
  Parent Trial Baseline Serostatus;Negative:Bivalent: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus;Negative:Bivalent | 14.0 [9.0 to 20.4] | 10.9 [3.6 to 23.6]
  Parent Trial Baseline Serostatus;Negative: Trivalent: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus;Negative: Trivalent | 21.7 [15.5 to 28.9] | 23.9 [12.6 to 38.8]
  Parent Trial Baseline Serostatus;Negative: Tetravalent: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus;Negative: Tetravalent | 56.1 [47.9 to 64.0] | 65.2 [49.8 to 78.6]

23. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. (DEN-304). All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 15 for parent trial DEN-304.
Time Frame: Month 15 (DEN-304)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304
Number analyzed (Participants) | 171
percentage of participants
  Parent Trial Baseline Serostatus; Positive: Bivalent: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus; Positive: Bivalent | 8.3 [1.0 to 27.0]
  Parent Trial Baseline Serostatus; Positive: Trivalent: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus; Positive: Trivalent | 8.3 [1.0 to 27.0]
  Parent Trial Baseline Serostatus; Positive: Tetravalent: number analyzed (Participants) | 24
  Parent Trial Baseline Serostatus; Positive: Tetravalent | 75.0 [53.3 to 90.2]
  Parent Trial Baseline Serostatus; Negative: Bivalent: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus; Negative: Bivalent | 10.9 [6.4 to 17.1]
  Parent Trial Baseline Serostatus; Negative: Trivalent: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus; Negative: Trivalent | 18.4 [12.5 to 25.6]
  Parent Trial Baseline Serostatus; Negative: Tetravalent: number analyzed (Participants) | 147
  Parent Trial Baseline Serostatus; Negative: Tetravalent | 68.0 [59.8 to 75.5]

24. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes in the Period Prior to Booster by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 42) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3 at Month 42 for parent trial DEN-315.
Time Frame: Month 42 (DEN-315)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior to Booster: DEN-315
Number analyzed (Participants) | 80
percentage of participants
  Parent Trial Baseline Serostatus; Positive: Bivalent: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus; Positive: Bivalent | 0 [0.0 to 41.0]
  Parent Trial Baseline Serostatus; Positive: Trivalent: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus; Positive: Trivalent | 42.9 [9.9 to 81.6]
  Parent Trial Baseline Serostatus; Positive: Tetravalent: number analyzed (Participants) | 7
  Parent Trial Baseline Serostatus; Positive: Tetravalent | 57.1 [18.4 to 90.1]
  Parent Trial Baseline Serostatus; Negative: Bivalent: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus; Negative: Bivalent | 21.9 [13.1 to 33.1]
  Parent Trial Baseline Serostatus; Negative: Trivalent: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus; Negative: Trivalent | 26.0 [16.5 to 37.6]
  Parent Trial Baseline Serostatus; Negative: Tetravalent: number analyzed (Participants) | 73
  Parent Trial Baseline Serostatus; Negative: Tetravalent | 47.9 [36.1 to 60.0]

25. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Pre-Booster Dose at Visit 3 for Both Parent Trials
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 3, pre-booster dose for all participants (Month 15 for parent trial DEN-304 and Month 42 for parent trial DEN-315). Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315)
Population: Per Protocol Set-Booster (PPS-B) included all participants from the FAS-B who received two doses of Takeda's TDV in the parent trials with no new major protocol violations after administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial. Overall number of participants analyzed: number of participants with data available for analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Booster Phase: Placebo: Participants received TDV placebo-matching 0.5 mL injection, subcutaneously, once at Visit 3 (Month 15) for participants from parent trial DEN-304 (US) or once at Visit 3 (Month 42) for participants from parent trial DEN-315 (Mexico).
- Booster Phase: TDV: Participants received TDV 0.5 mL, injection, subcutaneously, once at Visit 3 (Month 15) for participants from parent trials DEN-304 (US) or once at Visit 3 (Month 42) for participants from parent trial DEN-315 (Mexico).
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
titer
  DENV-1 | 116.2 [86.6 to 156.0] | 120.7 [86.9 to 167.8]
  DENV-2 | 404.0 [327.2 to 498.8] | 361.7 [279.7 to 467.9]
  DENV-3 | 32.3 [24.8 to 41.9] | 30.1 [22.5 to 40.3]
  DENV-4 | 20.8 [16.0 to 27.1] | 21.4 [16.1 to 28.3]

26. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 for Both Parent Trials
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 4, 1 month post-booster dose for all participants (Month 16 for parent trial DEN-304 and Month 43 for parent trial DEN-315).
Time Frame: 1 month post-booster dose at Month 16 (DEN-304) and Month 43 (DEN-315)
Population: PPS-B included all participants from the FAS-B who received two doses of Takeda's TDV in the parent trials with no new major protocol violations after administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial. Overall number of participants analyzed: number of participants with data available for analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 99 | 97
titer
  DENV-1 | 110.8 [82.2 to 149.5] | 1438.3 [1104.0 to 1873.8]
  DENV-2 | 363.4 [291.8 to 452.7] | 1038.8 [833.7 to 1294.4]
  DENV-3 | 27.7 [21.0 to 36.5] | 446.5 [356.8 to 558.8]
  DENV-4 | 20.0 [15.4 to 26.0] | 273.5 [213.2 to 350.8]

27. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Pre-Booster Dose at Visit 3 (Month 15) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the pre-booster data from Visit 3 at Month 15 for participants from parent trial DEN-304. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 61 | 61
titer
  DENV-1 | 126.4 [82.2 to 194.4] | 130.6 [81.9 to 208.4]
  DENV-2 | 583.9 [448.5 to 760.2] | 596.6 [453.4 to 785.1]
  DENV-3 | 36.9 [26.6 to 51.3] | 39.5 [26.3 to 59.6]
  DENV-4 | 31.3 [21.9 to 44.9] | 29.9 [19.9 to 44.8]

28. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 (Month 16) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 4 at Month 16 for participants from parent trial DEN-304.
Time Frame: 1 month post-booster dose at Month 16 (DEN-304)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 59 | 60
titer
  DENV-1 | 120.1 [78.5 to 184.0] | 1254.3 [862.2 to 1824.5]
  DENV-2 | 499.2 [379.7 to 656.4] | 1121.4 [867.5 to 1449.5]
  DENV-3 | 30.6 [21.4 to 43.5] | 389.7 [280.8 to 540.8]
  DENV-4 | 29.4 [20.5 to 42.2] | 260.9 [189.0 to 360.1]

29. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Pre-Booster Dose at Visit 3 (Month 42) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the pre-booster data from Visit 3 at Month 42 for participants from parent trial DEN-315. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 42 (DEN-315)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 41 | 39
titer
  DENV-1 | 102.6 [70.6 to 149.0] | 106.7 [68.3 to 166.7]
  DENV-2 | 233.5 [176.1 to 309.8] | 165.4 [110.7 to 247.1]
  DENV-3 | 26.4 [17.0 to 41.1] | 19.6 [13.6 to 28.2]
  DENV-4 | 11.3 [8.3 to 15.5] | 12.7 [9.4 to 17.1]

30. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 (Month 43) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 4 at Month 43 for participants from parent trial DEN-315.
Time Frame: 1 month post-booster dose at Month 43 (DEN-315)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 37
titer
  DENV-1 | 98.4 [65.1 to 148.7] | 1795.8 [1273.5 to 2532.5]
  DENV-2 | 227.5 [164.5 to 314.6] | 917.6 [607.2 to 1386.7]
  DENV-3 | 24.0 [15.2 to 37.8] | 556.8 [431.6 to 718.3]
  DENV-4 | 11.3 [8.3 to 15.4] | 295.3 [196.0 to 444.8]

31. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 for Both Parent Trials
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 3, pre-booster dose for all participants (Month 15 for parent trial DEN-304 and Month 42 for parent trial DEN-315). Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315)
Population: PPS-B included all participants from the FAS-B who received two doses of Takeda's TDV in the parent trials with no new major protocol violations after administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial. Overall number of participants analyzed: number of participants with data available for analyses. Number analyzed: number of participants with data available for analysis for the specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 165.0 [62.2 to 437.8] | 310.4 [67.2 to 1434.4]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 353.6 [192.1 to 650.8] | 771.3 [334.8 to 1776.9]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 53.8 [23.4 to 123.6] | 88.8 [25.1 to 313.4]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 27.7 [14.0 to 55.0] | 43.5 [10.6 to 177.6]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 110.4 [80.8 to 150.9] | 106.1 [77.2 to 145.9]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 411.9 [327.7 to 517.8] | 326.2 [249.4 to 426.7]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 30.0 [22.7 to 39.6] | 26.0 [19.6 to 34.4]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 20.0 [15.0 to 26.7] | 19.4 [14.8 to 25.4]

32. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 for Both Parent Trials
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 4, 1 month post-booster dose for all participants (Month 16 for parent trial DEN-304 and Month 43 for parent trial DEN-315).
Time Frame: 1 month post-booster dose at Month 16 (DEN-304) and Month 43 (DEN-315)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 99 | 97
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 170.5 [59.7 to 487.0] | 1192.5 [343.2 to 4143.7]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 264.2 [124.8 to 559.2] | 1533.3 [720.1 to 3264.5]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 46.2 [16.9 to 126.4] | 286.5 [124.6 to 658.9]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 34.4 [19.6 to 60.5] | 204.2 [83.4 to 500.1]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 104.4 [76.2 to 143.2] | 1473.2 [1129.4 to 1921.6]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 379.8 [301.1 to 479.0] | 988.3 [783.4 to 1246.9]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 25.8 [19.4 to 34.4] | 472.6 [374.1 to 597.1]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 18.6 [13.9 to 24.8] | 283.9 [218.3 to 369.2]

33. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 15) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the pre-booster data from Visit 3 at Month 15 for participants from parent trial DEN-304. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 61 | 61
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 120.5 [37.2 to 390.0] | 368.4 [44.6 to 3040.1]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 368.8 [175.4 to 775.7] | 839.4 [298.9 to 2357.3]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 39.4 [19.3 to 80.6] | 102.1 [19.0 to 549.3]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 22.9 [11.8 to 44.6] | 59.1 [10.3 to 339.8]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 127.6 [79.0 to 206.0] | 109.2 [70.2 to 169.7]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 639.0 [480.4 to 849.9] | 562.4 [423.1 to 747.5]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 36.4 [25.0 to 53.2] | 33.6 [22.5 to 50.1]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 33.3 [22.0 to 50.5] | 26.5 [17.8 to 39.5]

34. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 (Month 16) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 4 at Month 16 for participants from parent trial DEN-304.
Time Frame: 1 month post-booster dose at Month 16 (DEN-304)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 59 | 60
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 125.6 [32.3 to 488.7] | 1124.7 [182.3 to 6939.8]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 264.3 [105.0 to 665.2] | 1545.0 [528.1 to 4519.9]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 29.3 [11.6 to 74.3] | 239.1 [72.7 to 786.1]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 29.8 [19.5 to 45.6] | 202.8 [57.6 to 714.0]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 119.2 [75.0 to 189.3] | 1275.5 [879.5 to 1849.6]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 559.8 [422.3 to 742.0] | 1067.4 [820.0 to 1389.6]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 30.8 [20.7 to 45.8] | 420.1 [297.4 to 593.5]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 29.4 [19.2 to 44.8] | 271.1 [193.3 to 380.4]

35. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 42) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the pre-booster data from Visit 3 at Month 42 for participants from parent trial DEN-315. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 42 (DEN-315)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 41 | 39
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 470.4 [25.4 to 8709.7] | 185.7 [11.7 to 2940.9]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 307.1 [19.8 to 4754.2] | 598.4 [15.8 to 22694.8]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 151.1 [0.7 to 34960.6] | 58.2 [1.5 to 2257.4]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 52.5 [0.7 to 3894.5] | 17.2 [0.1 to 3545.3]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 91.0 [63.1 to 131.1] | 101.9 [63.5 to 163.5]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 228.5 [170.5 to 306.3] | 148.6 [99.7 to 221.4]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 23.0 [15.2 to 34.8] | 17.9 [12.5 to 25.7]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 10.0 [7.6 to 13.2] | 12.3 [9.4 to 16.2]

36. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 (Month 43) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 4 at Month 43 for participants from parent trial DEN-315.
Time Frame: 1 month post-booster dose at Month 43 (DEN-315)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 37
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 427.0 [45.4 to 4020.4] | 1393.8 [219.3 to 8859.8]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 264.1 [8.7 to 8032.8] | 1502.5 [236.0 to 9565.9]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 180.8 [1.1 to 29718.0] | 464.2 [204.7 to 1052.5]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 53.0 [0.9 to 3256.9] | 208.0 [18.4 to 2353.2]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 87.3 [57.6 to 132.5] | 1836.5 [1269.6 to 2656.5]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 224.8 [160.9 to 314.1] | 878.5 [563.9 to 1368.8]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 20.4 [13.4 to 31.0] | 565.8 [429.2 to 745.8]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 10.0 [7.7 to 13.1] | 304.5 [196.5 to 472.0]

37. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose at Visit 5 for Both Parent Trials
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 5, 6 months post-booster dose for all participants (Month 21 for parent trial DEN-304 and Month 48 for parent trial DEN-315).
Time Frame: 6 months post-booster dose at Month 21 (DEN-304) and Month 48 (DEN-315)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 96 | 92
titer
  DENV-1 | 94.2 [66.9 to 132.7] | 464.9 [336.1 to 642.9]
  DENV-2 | 305.2 [244.7 to 380.7] | 552.5 [442.1 to 690.5]
  DENV-3 | 27.4 [21.4 to 35.3] | 159.5 [122.6 to 207.4]
  DENV-4 | 16.7 [13.0 to 21.5] | 87.5 [65.8 to 116.2]

38. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose at Visit 5 (Month 21) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 5 at Month 21 for participants from parent trial DEN-304.
Time Frame: 6 months post-booster dose at Month 21 (DEN-304)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 56 | 54
titer
  DENV-1 | 107.8 [65.0 to 179.0] | 410.9 [259.7 to 650.1]
  DENV-2 | 433.0 [321.4 to 583.5] | 689.4 [530.6 to 895.8]
  DENV-3 | 30.7 [21.9 to 42.9] | 133.5 [90.5 to 197.0]
  DENV-4 | 24.3 [16.7 to 35.3] | 89.2 [60.5 to 131.7]

39. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose at Visit 5 (Month 48) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Reported here is the data from Visit 5 at Month 48 for participants from parent trial DEN-315.
Time Frame: 6 months post-booster dose at Month 48 (DEN-315)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 38
titer
  DENV-1 | 78.0 [50.6 to 120.2] | 553.9 [350.8 to 874.6]
  DENV-2 | 187.0 [142.3 to 245.6] | 403.4 [275.1 to 591.6]
  DENV-3 | 23.5 [15.9 to 34.6] | 205.2 [149.1 to 282.5]
  DENV-4 | 9.9 [7.8 to 12.5] | 85.0 [55.3 to 130.6]

40. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 for Both Parent Trials
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 5, 6 month post-booster dose for all participants (Month 21 for parent trial DEN-304 and Month 48 for parent trial DEN-315).
Time Frame: 6 months post-booster dose at Month 21 (DEN-304) and Month 48 (DEN-315)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 96 | 92
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 166.2 [48.3 to 571.7] | 435.8 [106.8 to 1777.8]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 278.9 [108.9 to 714.1] | 699.2 [305.0 to 1603.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 39.0 [18.8 to 80.8] | 137.1 [44.9 to 418.7]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 22.0 [12.1 to 40.1] | 83.6 [25.0 to 279.0]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 88.2 [61.5 to 126.5] | 469.4 [338.9 to 650.1]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 308.4 [245.1 to 387.9] | 533.4 [422.9 to 672.6]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 26.3 [20.1 to 34.5] | 163.1 [125.1 to 212.7]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 16.2 [12.3 to 21.3] | 88.1 [66.1 to 117.3]

41. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 (Month 21) (DEN-304)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 5 at Month 21 for participants from parent trial DEN-304.
Time Frame: 6 months post-booster dose at Month 21 (DEN-304)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 56 | 54
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 154.2 [30.2 to 786.6] | 461.7 [68.8 to 3098.9]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 337.6 [104.5 to 1090.2] | 825.4 [309.0 to 2205.1]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 37.5 [14.4 to 98.0] | 145.5 [32.0 to 661.2]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 21.7 [10.2 to 46.3] | 95.7 [21.6 to 423.2]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 101.6 [58.6 to 176.2] | 401.4 [254.9 to 632.2]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 451.4 [330.8 to 615.9] | 665.0 [508.0 to 870.6]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 29.7 [20.5 to 43.0] | 131.3 [88.3 to 195.1]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 24.8 [16.2 to 37.9] | 88.0 [59.0 to 131.2]

42. Primary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 (Month 48) (DEN-315)
Description: GMTs of neutralizing antibodies were measured by MNT50 for each of the 4 Dengue Serotypes (DENV-1, DENV-2, DENV-3 and DENV-4). Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. Reported here is the data from Visit 5 at Month 48 for participants from parent trial DEN-315.
Time Frame: 6 months post-booster dose at Month 48 (DEN-315)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 38
titer
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 223.9 [31.8 to 1574.3] | 366.4 [8.2 to 16297.5]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 129.9 [0.8 to 21199.9] | 425.0 [9.5 to 19098.8]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 45.5 [6.5 to 319.1] | 114.5 [6.0 to 2196.9]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 23.2 [0.0 to 23073.9] | 55.8 [0.3 to 10826.4]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 73.8 [47.1 to 115.6] | 573.9 [355.3 to 927.0]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 190.6 [143.4 to 253.4] | 401.6 [269.9 to 597.6]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 22.7 [15.1 to 34.0] | 215.7 [155.4 to 299.5]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 9.4 [7.5 to 11.9] | 88.2 [57.3 to 135.7]

43. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at Pre-Booster Dose at Visit 3 for Both Parent Trials
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3, pre-booster dose for all participants (Month 15 for parent trial DEN-304 and Month 42 for parent trial DEN-315). Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Booster Phase: Placebo: Participants received TDV placebo-matching 0.5 ml injection, SC, once at Visit 3 (Month 15) for participants from parent trial DEN-304 (US) or once at Visit 3 (Month 42) for participants from parent trial DEN-315 (Mexico).
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
percentage of participants
  DENV-1 | 98.0 [93.1 to 99.8] | 94.0 [87.4 to 97.8]
  DENV-2 | 100 [96.4 to 100.0] | 99.0 [94.6 to 100.0]
  DENV-3 | 80.4 [71.4 to 87.6] | 73.0 [63.2 to 81.4]
  DENV-4 | 66.7 [56.6 to 75.7] | 67.0 [56.9 to 76.1]

44. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 for Both Parent Trials
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4, 1 month post-booster dose for all participants (Month 16 for parent trial DEN-304 and Month 43 for parent trial DEN-315).
Time Frame: 1 month post-booster dose at Month 16 (DEN-304) and Month 43 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 99 | 97
percentage of participants
  DENV-1 | 98.0 [92.9 to 99.8] | 100 [96.3 to 100.0]
  DENV-2 | 100 [96.3 to 100.0] | 100 [96.3 to 100.0]
  DENV-3 | 71.7 [61.8 to 80.3] | 100 [96.3 to 100.0]
  DENV-4 | 66.7 [56.5 to 75.8] | 100 [96.3 to 100.0]

45. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at Pre-Booster Dose at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 15 for participants from parent trial DEN-304. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 61 | 61
percentage of participants
  DENV-1 | 96.7 [88.7 to 99.6] | 95.1 [86.3 to 99.0]
  DENV-2 | 100 [94.1 to 100.0] | 100 [94.1 to 100.0]
  DENV-3 | 83.6 [71.9 to 91.8] | 77.0 [64.5 to 86.8]
  DENV-4 | 75.4 [62.7 to 85.5] | 72.1 [59.2 to 82.9]

46. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 (Month 16) (DEN-304)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 16 for participants from parent trial DEN-304.
Time Frame: 1 month post-booster dose at Month 16 (DEN-304)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 59 | 60
percentage of participants
  DENV-1 | 98.3 [90.9 to 100.0] | 100 [94.0 to 100.0]
  DENV-2 | 100 [93.9 to 100.0] | 100 [94.0 to 100.0]
  DENV-3 | 74.6 [61.6 to 85.0] | 100 [94.0 to 100.0]
  DENV-4 | 76.3 [63.4 to 86.4] | 100 [94.0 to 100.0]

47. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at Pre-Booster Dose at Visit 3 (Month 42) (DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 42 for participants from parent trial DEN-315. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 42 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 41 | 39
percentage of participants
  DENV-1 | 100 [91.4 to 100.0] | 92.3 [79.1 to 98.4]
  DENV-2 | 100 [91.4 to 100.0] | 97.4 [86.5 to 99.9]
  DENV-3 | 75.6 [59.7 to 87.6] | 66.7 [49.8 to 80.9]
  DENV-4 | 53.7 [37.4 to 69.3] | 59.0 [42.1 to 74.4]

48. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 (Month 43) (DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 43 for participants from parent trial DEN-315.
Time Frame: 1 month post-booster dose at Month 43 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 37
percentage of participants
  DENV-1 | 97.5 [86.8 to 99.9] | 100 [90.5 to 100.0]
  DENV-2 | 100 [91.2 to 100.0] | 100 [90.5 to 100.0]
  DENV-3 | 67.5 [50.9 to 81.4] | 100 [90.5 to 100.0]
  DENV-4 | 52.5 [36.1 to 68.5] | 100 [90.5 to 100.0]

49. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 for Both Parent Trials
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3, pre-booster dose for all participants (Month 15 for parent trial DEN-304 and Month 42 for parent trial DEN-315). Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 92.3 [64.0 to 99.8] | 91.7 [61.5 to 99.8]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [75.3 to 100.0] | 100 [73.5 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 92.3 [64.0 to 99.8] | 83.3 [51.6 to 97.9]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 84.6 [54.6 to 98.1] | 66.7 [34.9 to 90.1]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 98.9 [93.9 to 100.0] | 94.3 [87.2 to 98.1]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [95.9 to 100.0] | 98.9 [93.8 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 78.7 [68.7 to 86.6] | 71.6 [61.0 to 80.7]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 64.0 [53.2 to 73.9] | 67.0 [56.2 to 76.7]

50. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 for Both Parent Trials
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4, 1 month post-booster dose for all participants (Month 16 for parent trial DEN-304 and Month 43 for parent trial DEN-315).
Time Frame: 1 month post-booster dose at Month 16 (DEN-304) and Month 43 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 99 | 97
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 91.7 [61.5 to 99.8] | 100 [71.5 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [73.5 to 100.0] | 100 [71.5 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 83.3 [51.6 to 97.9] | 100 [71.5 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 100 [73.5 to 100.0] | 100 [71.5 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 98.9 [93.8 to 100.0] | 100 [95.8 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [95.8 to 100.0] | 100 [95.8 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 70.1 [59.4 to 79.5] | 100 [95.8 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 62.1 [51.0 to 72.3] | 100 [95.8 to 100.0]

51. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 15 for participants from parent trial DEN-304. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 61 | 61
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 90.0 [55.5 to 99.7] | 88.9 [51.8 to 99.7]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [69.2 to 100.0] | 100 [66.4 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 90.0 [55.5 to 99.7] | 77.8 [40.0 to 97.2]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 80.0 [44.4 to 97.5] | 77.8 [40.0 to 97.2]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 98.0 [89.6 to 100.0] | 96.2 [86.8 to 99.5]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [93.0 to 100.0] | 100 [93.2 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 82.4 [69.1 to 91.6] | 76.9 [63.2 to 87.5]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 74.5 [60.4 to 85.7] | 71.2 [56.9 to 82.9]

52. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 (Month 16) (DEN-304)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 16 for participants from parent trial DEN-304.
Time Frame: 1 month post-booster dose at Month 16 (DEN-304)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 59 | 60
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 88.9 [51.8 to 99.7] | 100 [63.1 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [66.4 to 100.0] | 100 [63.1 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 77.8 [40.0 to 97.2] | 100 [63.1 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 100 [66.4 to 100.0] | 100 [63.1 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 100 [92.9 to 100.0] | 100 [93.2 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [92.9 to 100.0] | 100 [93.2 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 74.0 [59.7 to 85.4] | 100 [93.2 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 72.0 [57.5 to 83.8] | 100 [93.2 to 100.0]

53. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 42) (DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 42 for participants from parent trial DEN-315. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 42 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 41 | 39
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 3 | 39
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 100 [29.2 to 100.0] | 33.3 [0.8 to 90.6]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 100 [90.7 to 100.0] | 91.7 [77.5 to 98.2]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [90.7 to 100.0] | 97.2 [85.5 to 99.9]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 73.7 [56.9 to 86.6] | 63.9 [46.2 to 79.2]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 50.0 [33.4 to 66.6] | 61.1 [43.5 to 76.9]

54. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 (Month 43) (DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 43 for participants from parent trial DEN-315.
Time Frame: 1 month post-booster dose at Month 43 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 37
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 97.3 [85.8 to 99.9] | 100 [89.7 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [90.5 to 100.0] | 100 [89.7 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 64.9 [47.5 to 79.8] | 100 [89.7 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 48.6 [31.9 to 65.6] | 100 [89.7 to 100.0]

55. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose at Visit 5 for Both Parent Trials
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5, 6 month post-booster dose for all participants (Month 21 for parent trial DEN-304 and Month 48 for parent trial DEN-315).
Time Frame: 6 months post-booster dose at Month 21 (DEN-304) and Month 48 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 96 | 92
percentage of participants
  DENV-1 | 90.6 [82.9 to 95.6] | 96.7 [90.8 to 99.3]
  DENV-2 | 100 [96.2 to 100.0] | 100 [96.1 to 100.0]
  DENV-3 | 76.0 [66.3 to 84.2] | 98.9 [94.1 to 100.0]
  DENV-4 | 63.5 [53.1 to 73.1] | 94.6 [87.8 to 98.2]

56. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose at Visit 5 (Month 21) (DEN-304)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 21 for participants from parent trial DEN-304.
Time Frame: 6 months post-booster dose at Month 21 (DEN-304)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 56 | 54
percentage of participants
  DENV-1 | 89.3 [78.1 to 96.0] | 96.3 [87.3 to 99.5]
  DENV-2 | 100 [93.6 to 100.0] | 100 [93.4 to 100.0]
  DENV-3 | 78.6 [65.6 to 88.4] | 98.1 [90.1 to 100.0]
  DENV-4 | 71.4 [57.8 to 82.7] | 96.3 [87.3 to 99.5]

57. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose at Visit 5 (Month 48) (DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 48 for participants from parent trial DEN-315.
Time Frame: 6 months post-booster dose at Month 48 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 38
percentage of participants
  DENV-1 | 92.5 [79.6 to 98.4] | 97.4 [86.2 to 99.9]
  DENV-2 | 100 [91.2 to 100.0] | 100 [90.7 to 100.0]
  DENV-3 | 72.5 [56.1 to 85.4] | 100 [90.7 to 100.0]
  DENV-4 | 52.5 [36.1 to 68.5] | 92.1 [78.6 to 98.3]

58. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 for Both Parent Trials
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5, 6 month post-booster dose for all participants (Month 21 for parent trial DEN-304 and Month 48 for parent trial DEN-315).
Time Frame: 6 months post-booster dose at Month 21 (DEN-304) and Month 48 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 96 | 92
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 90.0 [55.5 to 99.7] | 91.7 [61.5 to 99.8]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [69.2 to 100.0] | 100 [73.5 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 90.0 [55.5 to 99.7] | 91.7 [61.5 to 99.8]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 90.0 [55.5 to 99.7] | 83.3 [51.6 to 97.9]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 90.7 [82.5 to 95.9] | 97.5 [91.3 to 99.7]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [95.8 to 100.0] | 100 [95.5 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 74.4 [63.9 to 83.2] | 100 [95.5 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 60.5 [49.3 to 70.8] | 96.3 [89.4 to 99.2]

59. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 (Month 21) (DEN-304)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 21 for participants from parent trial DEN-304.
Time Frame: 6 months post-booster dose at Month 21 (DEN-304)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 56 | 54
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 87.5 [47.3 to 99.7] | 88.9 [51.8 to 99.7]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [63.1 to 100.0] | 100 [66.4 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 87.5 [47.3 to 99.7] | 88.9 [51.8 to 99.7]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 87.5 [47.3 to 99.7] | 88.9 [51.8 to 99.7]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 89.6 [77.3 to 96.5] | 97.8 [88.2 to 99.9]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [92.6 to 100.0] | 100 [92.1 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 77.1 [62.7 to 88.0] | 100 [92.1 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 68.8 [53.7 to 81.3] | 97.8 [88.2 to 99.9]

60. Primary Outcome: Seropositivity Rate for Each of the 4 Dengue Serotypes at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 (Month 48) (DEN-315)
Description: Seropositivity rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 48 for participants from parent trial DEN-315.
Time Frame: 6 months post-booster dose at Month 48 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 38
percentage of participants
  Parent Trial Baseline Serostatus;Positive: DENV-1: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-1 | 100 [15.8 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-2: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-2 | 100 [15.8 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-3: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-3 | 100 [15.8 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus;Positive: DENV-4: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus;Positive: DENV-4 | 100 [15.8 to 100.0] | 66.7 [9.4 to 99.2]
  Parent Trial Baseline Serostatus;Negative: DENV-1: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-1 | 92.1 [78.6 to 98.3] | 97.1 [85.1 to 99.9]
  Parent Trial Baseline Serostatus;Negative: DENV-2: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-2 | 100 [90.7 to 100.0] | 100 [90.0 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-3: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-3 | 71.1 [54.1 to 84.6] | 100 [90.0 to 100.0]
  Parent Trial Baseline Serostatus;Negative: DENV-4: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus;Negative: DENV-4 | 50.0 [33.4 to 66.6] | 94.3 [80.8 to 99.3]

61. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at Pre-Booster Dose at Visit 3 for Both Parent Trials
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3, pre-booster dose for all participants (Month 15 for parent trial DEN-304 and Month 42 for parent trial DEN-315). Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
percentage of participants
  Bivalent | 15.7 [9.2 to 24.2] | 16.0 [9.4 to 24.7]
  Trivalent | 20.6 [13.2 to 29.7] | 20.0 [12.7 to 29.2]
  Tetravalent | 62.7 [52.6 to 72.1] | 59.0 [48.7 to 68.7]

62. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 for Both Parent Trials
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4, 1 month post-booster dose for all participants (Month 16 for parent trial DEN-304 and Month 43 for parent trial DEN-315).
Time Frame: 1 month post-booster dose at Month 16 (DEN-304) and Month 43 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 99 | 97
percentage of participants
  Bivalent | 18.2 [11.1 to 27.2] | 0 [0.0 to 3.7]
  Trivalent | 24.2 [16.2 to 33.9] | 0 [0.0 to 3.7]
  Tetravalent | 56.6 [46.2 to 66.5] | 100 [96.3 to 100.0]

63. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at Pre-Booster Dose at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 15 for participants from parent trial DEN-304. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 61 | 61
percentage of participants
  Bivalent | 11.5 [4.7 to 22.2] | 14.8 [7.0 to 26.2]
  Trivalent | 16.4 [8.2 to 28.1] | 16.4 [8.2 to 28.1]
  Tetravalent | 70.5 [57.4 to 81.5] | 65.6 [52.3 to 77.3]

64. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at 1 Month Post-Booster Dose at Visit 4 (Month 16) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 16 for participants from parent trial DEN-304.
Time Frame: 1 month post-booster dose at Month 16 (DEN-304.)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 59 | 60
percentage of participants
  Bivalent | 15.3 [7.2 to 27.0] | 0 [0.0 to 6.0]
  Trivalent | 20.3 [11.0 to 32.8] | 0 [0.0 to 6.0]
  Tetravalent | 64.4 [50.9 to 76.4] | 100 [94.0 to 100.0]

65. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at Pre-Booster Dose at Visit 3 (Month 42) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 42 for participants from parent trial DEN-315. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 42 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 41 | 39
percentage of participants
  Bivalent | 22.0 [10.6 to 37.6] | 17.9 [7.5 to 33.5]
  Trivalent | 26.8 [14.2 to 42.9] | 25.6 [13.0 to 42.1]
  Tetravalent | 51.2 [35.1 to 67.1] | 48.7 [32.4 to 65.2]

66. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes Post-Booster Dose at 1 Month Post-Booster Dose at Visit 4 (Month 43) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 43 for participants from parent trial DEN-315.
Time Frame: 1 month post-booster dose at Month 43 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 37
percentage of participants
  Bivalent | 22.5 [10.8 to 38.5] | 0 [0.0 to 9.5]
  Trivalent | 30.0 [16.6 to 46.5] | 0 [0.0 to 9.5]
  Tetravalent | 45.0 [29.3 to 61.5] | 100 [90.5 to 100.0]

67. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 for Both Parent Trials
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), \ any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 3, pre-booster dose for all participants (Month 15 for parent trial DEN-304 and Month 42 for parent trial DEN-315). Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus: Positive; Bivalent | 7.7 [0.2 to 36.0] | 8.3 [0.2 to 38.5]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus: Positive; Trivalent | 15.4 [1.9 to 45.4] | 16.7 [2.1 to 48.4]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 13 | 12
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 76.9 [46.2 to 95.0] | 66.7 [34.9 to 90.1]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus: Negative; Bivalent | 16.9 [9.8 to 26.3] | 17.0 [9.9 to 26.6]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus: Negative; Trivalent | 21.3 [13.4 to 31.3] | 20.5 [12.6 to 30.4]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 89 | 88
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 60.7 [49.7 to 70.9] | 58.0 [47.0 to 68.4]

68. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 for Both Parent Trials
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), \ any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4, 1 month post-booster dose for all participants (Month 16 for parent trial DEN-304 and Month 43 for parent trial DEN-315).
Time Frame: 1 month post-booster dose at Month 16 (DEN-304) and Month 43 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 99 | 97
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Bivalent | 8.3 [0.2 to 38.5] | 0 [0.0 to 28.5]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Trivalent | 8.3 [0.2 to 38.5] | 0 [0.0 to 28.5]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 83.3 [51.6 to 97.9] | 100 [71.5 to 100.0]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus: Negative; Bivalent | 19.5 [11.8 to 29.4] | 0 [0.0 to 4.2]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus: Negative; Trivalent | 26.4 [17.6 to 37.0] | 0 [0.0 to 4.2]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 52.9 [41.9 to 63.7] | 100 [95.8 to 100.0]

69. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 15) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), \ any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 15 for participants from parent trial DEN-304. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 15 (DEN-304)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 61 | 61
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus: Positive; Bivalent | 10.0 [0.3 to 44.5] | 11.1 [0.3 to 48.2]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus: Positive; Trivalent | 20.0 [2.5 to 55.6] | 0 [0.0 to 33.6]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 10 | 9
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 70.0 [34.8 to 93.3] | 77.8 [40.0 to 97.2]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus: Negative; Bivalent | 11.8 [4.4 to 23.9] | 15.4 [6.9 to 28.1]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus: Negative; Trivalent | 15.7 [7.0 to 28.6] | 19.2 [9.6 to 32.5]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 51 | 52
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 70.6 [56.2 to 82.5] | 63.5 [49.0 to 76.4]

70. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 (Month 16) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), \any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 16 for participants from parent trial DEN-304.
Time Frame: 1 month post-booster dose at Month 16 (DEN-304)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 59 | 60
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus: Positive; Bivalent | 11.1 [0.3 to 48.2] | 0 [0.0 to 36.9]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus: Positive; Trivalent | 11.1 [0.3 to 48.2] | 0 [0.0 to 36.9]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 9 | 8
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 77.8 [40.0 to 97.2] | 100 [63.1 to 100.0]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus: Negative; Bivalent | 16.0 [7.2 to 29.1] | 0 [0.0 to 6.8]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus: Negative; Trivalent | 22.0 [11.5 to 36.0] | 0 [0.0 to 6.8]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 50 | 52
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 62.0 [47.2 to 75.3] | 100 [93.2 to 100.0]

71. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at Pre-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 3 (Month 42) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the pre-booster data from Visit 3 at Month 42 for participants from parent trial DEN-315. Pre-booster dose is defined as the last non-missing value before booster administration.
Time Frame: Pre-booster dose at Month 42 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 41 | 39
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus: Positive; Bivalent | 0 [0.0 to 70.8] | 0 [0.0 to 70.8]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus: Positive; Trivalent | 0 [0.0 to 70.8] | 66.7 [9.4 to 99.2]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 100 [29.2 to 100.0] | 33.3 [0.8 to 90.6]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus: Negative; Bivalent | 23.7 [11.4 to 40.2] | 19.4 [8.2 to 36.0]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus: Negative; Trivalent | 28.9 [15.4 to 45.9] | 22.2 [10.1 to 39.2]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 38 | 36
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 47.4 [31.0 to 64.2] | 50.0 [32.9 to 67.1]

72. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes at 1 Month Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 4 (Month 43) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 4 at Month 43 for participants from parent trial DEN-315.
Time Frame: 1 month post-booster dose at Month 43 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 37
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus: Positive; Bivalent | 0 [0.0 to 70.8] | 0 [0.0 to 70.8]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus: Positive; Trivalent | 0 [0.0 to 70.8] | 0 [0.0 to 70.8]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 3 | 3
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 100 [29.2 to 100.0] | 100 [29.2 to 100.0]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus: Negative; Bivalent | 24.3 [11.8 to 41.2] | 0 [0.0 to 10.3]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus: Negative; Trivalent | 32.4 [18.0 to 49.8] | 0 [0.0 to 10.3]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 37 | 34
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 40.5 [24.8 to 57.9] | 100 [89.7 to 100.0]

73. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes Post-Booster Dose at 6 Months Post-Booster Dose at Visit 5 for Both Parent Trials
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5, 6 month post-booster dose for all participants (Month 21 for parent trial DEN-304 and Month 48 for parent trial DEN-315).
Time Frame: 6 months post-booster dose at Month 21 (DEN-304) and Month 48 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 96 | 92
percentage of participants
  Bivalent | 14.6 [8.2 to 23.3] | 2.2 [0.3 to 7.6]
  Trivalent | 21.9 [14.1 to 31.5] | 5.4 [1.8 to 12.2]
  Tetravalent | 57.3 [46.8 to 67.3] | 92.4 [84.9 to 96.9]

74. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes Post-Booster Dose at 6 Months Post-Booster Dose at Visit 5 (Month 21) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 21 for participants from parent trial DEN-304.
Time Frame: 6 months post-booster dose at Month 21 (DEN-304)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 56 | 54
percentage of participants
  Bivalent | 14.3 [6.4 to 26.2] | 1.9 [0.0 to 9.9]
  Trivalent | 16.1 [7.6 to 28.3] | 5.6 [1.2 to 15.4]
  Tetravalent | 64.3 [50.4 to 76.6] | 92.6 [82.1 to 97.9]

75. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes Post-booster Dose at 6 Months Post-Booster Dose at Visit 5 (Month 48) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 48 for participants from parent trial DEN-315.
Time Frame: 6 months post-Booster dose at Month 48 (DEN-315)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 38
percentage of participants
  Bivalent | 15.0 [5.7 to 29.8] | 2.6 [0.1 to 13.8]
  Trivalent | 30.0 [16.6 to 46.5] | 5.3 [0.6 to 17.7]
  Tetravalent | 47.5 [31.5 to 63.9] | 92.1 [78.6 to 98.3]

76. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes Post-Booster Dose at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 for Both Parent Trials
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5, 6 month post-booster dose for all participants (Month 21 for parent trial DEN-304 and Month 48 for parent trial DEN-315).
Time Frame: 6 months post-booster dose at Month 21 (DEN-304) and Month 48 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 96 | 92
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Bivalent | 0 [0.0 to 30.8] | 8.3 [0.2 to 38.5]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Trivalent | 0 [0.0 to 30.8] | 16.7 [2.1 to 48.4]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 90.0 [55.5 to 99.7] | 75.0 [42.8 to 94.5]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus: Negative; Bivalent | 16.3 [9.2 to 25.8] | 1.3 [0.0 to 6.8]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus: Negative; Trivalent | 24.4 [15.8 to 34.9] | 3.8 [0.8 to 10.6]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 53.5 [42.4 to 64.3] | 95.0 [87.7 to 98.6]

77. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes Post-Booster Dose at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 (Month 21) (DEN-304)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 21 for participants from parent trial DEN-304.
Time Frame: 6 months post-booster dose at Month 21 (DEN-304)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 56 | 54
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus: Positive; Bivalent | 0 [0.0 to 36.9] | 11.1 [0.3 to 48.2]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus: Positive; Trivalent | 0 [0.0 to 36.9] | 11.1 [0.3 to 48.2]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 8 | 9
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 87.5 [47.3 to 99.7] | 77.8 [40.0 to 97.2]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus: Negative; Bivalent | 16.7 [7.5 to 30.2] | 0 [0.0 to 7.9]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus: Negative; Trivalent | 18.8 [8.9 to 32.6] | 4.4 [0.5 to 15.1]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 48 | 45
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 60.4 [45.3 to 74.2] | 95.6 [84.9 to 99.5]

78. Primary Outcome: Seropositivity Rate for Multiple (2, 3 or 4) Dengue Serotypes Post-booster Dose at 6 Months Post-Booster Dose by Serostatus at Baseline in the Parent Trials at Visit 5 (Month 48) (DEN-315)
Description: Seropositivity rate for multiple Dengue serotypes, defined as the percentage of participants seropositive for more than one Dengue serotype, is derived from the titers of dengue-neutralizing antibodies. All 4 dengue serotypes (tetravalent), any 2 of the 4 dengue serotypes (bivalent), any 3 of the 4 dengue serotypes (trivalent). Seropositivity is defined as a reciprocal neutralizing titer ≥10. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Reported here is the data from Visit 5 at Month 48 for participants from parent trial DEN-315.
Time Frame: 6 months post-Booster dose at Month 48 (DEN-315)
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 40 | 38
percentage of participants
  Parent Trial Baseline Serostatus: Positive; Bivalent: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus: Positive; Bivalent | 0 [0.0 to 84.2] | 0 [0.0 to 70.8]
  Parent Trial Baseline Serostatus: Positive; Trivalent: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus: Positive; Trivalent | 0 [0.0 to 84.2] | 33.3 [0.8 to 90.6]
  Parent Trial Baseline Serostatus: Positive; Tetravalent: number analyzed (Participants) | 2 | 3
  Parent Trial Baseline Serostatus: Positive; Tetravalent | 100 [15.8 to 100.0] | 66.7 [9.4 to 99.2]
  Parent Trial Baseline Serostatus: Negative; Bivalent: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus: Negative; Bivalent | 15.8 [6.0 to 31.3] | 2.9 [0.1 to 14.9]
  Parent Trial Baseline Serostatus: Negative; Trivalent: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus: Negative; Trivalent | 31.6 [17.5 to 48.7] | 2.9 [0.1 to 14.9]
  Parent Trial Baseline Serostatus: Negative; Tetravalent: number analyzed (Participants) | 38 | 35
  Parent Trial Baseline Serostatus: Negative; Tetravalent | 44.7 [28.6 to 61.7] | 94.3 [80.8 to 99.3]

79. Secondary Outcome: Geometric Mean Ratio (GMR) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes for All Participants Prior to the Booster Dose
Description: The geometric mean ratio is the geometric mean of the ratio of the two visits being compared.
Time Frame: Month 12 vs Month 0, Month 15 (DEN-304) vs parent trial Month 4, Mont 42 (DEN315) vs parent trial Month 4, Month 0 vs parent trial Month 9, Month 12 vs parent trial Month 9
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
unitless ratio
  Month 12 vs Month 0: DENV-1: number analyzed (Participants) | 182 | 48
  Month 12 vs Month 0: DENV-1 | 0.753 [0.675 to 0.840] | 0.891 [0.741 to 1.071]
  Month 12 vs Month 0: DENV-2: number analyzed (Participants) | 182 | 48
  Month 12 vs Month 0: DENV-2 | 0.698 [0.650 to 0.749] | 0.622 [0.548 to 0.705]
  Month 12 vs Month 0: DENV-3: number analyzed (Participants) | 182 | 48
  Month 12 vs Month 0: DENV-3 | 0.864 [0.791 to 0.945] | 0.852 [0.668 to 1.088]
  Month 12 vs Month 0: DENV-4: number analyzed (Participants) | 182 | 48
  Month 12 vs Month 0: DENV-4 | 0.689 [0.632 to 0.751] | 0.861 [0.708 to 1.046]
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 167 | 0
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-1 | 0.438 [0.382 to 0.502] |
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 167 | 0
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-2 | 0.159 [0.137 to 0.185] |
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-3: number analyzed (Participants) | 167 | 0
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-3 | 0.275 [0.241 to 0.315] |
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 167 | 0
  Month 15 (DEN-304) vs Parent Trial Month 4: DENV-4 | 0.216 [0.183 to 0.255] |
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 0 | 73
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-1 |  | 0.296 [0.240 to 0.366]
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 0 | 73
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-2 |  | 0.108 [0.089 to 0.130]
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-3: number analyzed (Participants) | 0 | 73
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-3 |  | 0.202 [0.162 to 0.252]
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 0 | 73
  Month 42 (DEN-315) vs Parent Trial Month 4: DENV-4 |  | 0.066 [0.055 to 0.079]
  Month 0 vs Parent Trial Month 9: DENV-1: number analyzed (Participants) | 234 | 110
  Month 0 vs Parent Trial Month 9: DENV-1 | 0.529 [0.482 to 0.582] | 0.517 [0.455 to 0.587]
  Month 0 vs Parent Trial Month 9: DENV-2: number analyzed (Participants) | 234 | 110
  Month 0 vs Parent Trial Month 9: DENV-2 | 0.396 [0.369 to 0.426] | 0.466 [0.415 to 0.522]
  Month 0 vs Parent Trial Month 9: DENV-3: number analyzed (Participants) | 234 | 110
  Month 0 vs Parent Trial Month 9: DENV-3 | 0.440 [0.394 to 0.492] | 0.547 [0.477 to 0.629]
  Month 0 vs Parent Trial Month 9: DENV-4: number analyzed (Participants) | 234 | 110
  Month 0 vs Parent Trial Month 9: DENV-4 | 0.577 [0.518 to 0.641] | 0.568 [0.504 to 0.641]
  Month 12 vs Parent Trial Month 9: DENV-1: number analyzed (Participants) | 179 | 45
  Month 12 vs Parent Trial Month 9: DENV-1 | 0.415 [0.367 to 0.470] | 0.486 [0.377 to 0.627]
  Month 12 vs Parent Trial Month 9: DENV-2: number analyzed (Participants) | 179 | 45
  Month 12 vs Parent Trial Month 9: DENV-2 | 0.265 [0.239 to 0.295] | 0.289 [0.238 to 0.351]
  Month 12 vs Parent Trial Month 9: DENV-3: number analyzed (Participants) | 179 | 45
  Month 12 vs Parent Trial Month 9: DENV-3 | 0.407 [0.353 to 0.470] | 0.435 [0.336 to 0.562]
  Month 12 vs Parent Trial Month 9: DENV-4: number analyzed (Participants) | 179 | 45
  Month 12 vs Parent Trial Month 9: DENV-4 | 0.384 [0.335 to 0.440] | 0.567 [0.431 to 0.745]

80. Secondary Outcome: Geometric Mean Ratio (GMR) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes by Serostatus at Baseline in the Parent Trials Prior to the Booster Dose
Description: The geometric mean ratio is the geometric mean of the ratio of the two visits being compared. Baseline seropositivity is defined as reciprocal neutralizing titer ≥10 for one or more dengue serotypes at baseline in the parent trial.
Time Frame: Month 12 vs Month 0, Month 15 (DEN-304) vs parent trial Month 4, Month 42 (DEN315) vs parent trial Month 4, Month 0 vs parent trial Month 9, Month 12 vs parent trial Month 9
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 239 | 119
unitless ratio
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-1: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-1 | 0.736 [0.556 to 0.974] | 0.705 [0.002 to 222.445]
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-2: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-2 | 0.756 [0.599 to 0.955] | 0.456 [0.056 to 3.733]
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-3: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-3 | 0.980 [0.834 to 1.152] | 1.000 [NA to NA] — The confidence interval was not estimable due to an observed standard deviation of 0.
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-4: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Month 0: DENV-4 | 0.736 [0.598 to 0.906] | 0.727 [0.064 to 8.280]
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 24 | 0
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-1 | 0.506 [0.349 to 0.733] |
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 24 | 0
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-2 | 0.164 [0.108 to 0.249] |
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-3: number analyzed (Participants) | 24 | 0
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-3 | 0.350 [0.238 to 0.514] |
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 24 | 0
  Parent Trial Baseline Serostatus: Positive; Month 15 (DEN-304) vs Parent Trial Month 4: DENV-4 | 0.178 [0.125 to 0.253] |
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 0 | 7
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-1 |  | 0.393 [0.155 to 0.998]
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 0 | 7
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-2 |  | 0.164 [0.066 to 0.408]
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-3: number analyzed (Participants) | 0 | 7
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-3 |  | 0.319 [0.204 to 0.499]
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 0 | 7
  Parent Trial Baseline Serostatus: Positive; Month 42 (DEN-315) vs Parent Trial Month 4: DENV-4 |  | 0.070 [0.036 to 0.138]
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-1: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-1 | 0.635 [0.467 to 0.864] | 0.528 [0.453 to 0.616]
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-2: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-2 | 0.469 [0.356 to 0.619] | 0.454 [0.312 to 0.661]
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-3: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-3 | 0.538 [0.361 to 0.801] | 0.556 [0.356 to 0.868]
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-4: number analyzed (Participants) | 33 | 8
  Parent Trial Baseline Serostatus: Positive; Month 0 vs Parent Trial Month 9: DENV-4 | 0.710 [0.475 to 1.062] | 0.684 [0.401 to 1.165]
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-1: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-1 | 0.497 [0.330 to 0.748] | 0.375 [0.000 to 400.159]
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-2: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-2 | 0.311 [0.203 to 0.477] | 0.172 [0.161 to 0.184]
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-3: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-3 | 0.561 [0.329 to 0.957] | 0.664 [0.004 to 119.652]
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-4: number analyzed (Participants) | 25 | 2
  Parent Trial Baseline Serostatus: Positive; Month 12 vs Parent Trial Month 9: DENV-4 | 0.577 [0.335 to 0.994] | 0.966 [0.005 to 194.455]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-1: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-1 | 0.756 [0.671 to 0.851] | 0.900 [0.745 to 1.088]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-2: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-2 | 0.689 [0.639 to 0.742] | 0.630 [0.553 to 0.718]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-3: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-3 | 0.847 [0.767 to 0.936] | 0.846 [0.656 to 1.092]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-4: number analyzed (Participants) | 157 | 46
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Month 0; DENV-4 | 0.681 [0.619 to 0.750] | 0.867 [0.708 to 1.063]
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-1: number analyzed (Participants) | 143 | 0
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-1 | 0.427 [0.368 to 0.496] |
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-2: number analyzed (Participants) | 143 | 0
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-2 | 0.158 [0.135 to 0.186] |
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-3: number analyzed (Participants) | 143 | 0
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-3 | 0.265 [0.229 to 0.305] |
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-4: number analyzed (Participants) | 143 | 0
  Parent Trial Baseline Serostatus: Negative; Month 15 (DEN-304) vs Parent Trial Month 4; DENV-4 | 0.223 [0.186 to 0.268] |
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-1: number analyzed (Participants) | 0 | 66
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-1 |  | 0.288 [0.231 to 0.359]
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-2: number analyzed (Participants) | 0 | 66
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-2 |  | 0.103 [0.085 to 0.125]
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-3: number analyzed (Participants) | 0 | 66
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-3 |  | 0.192 [0.152 to 0.244]
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-4: number analyzed (Participants) | 0 | 66
  Parent Trial Baseline Serostatus: Negative; Month 42 (DEN-315) vs Parent Trial Month 4; DENV-4 |  | 0.065 [0.053 to 0.080]
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-1: number analyzed (Participants) | 201 | 102
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-1 | 0.514 [0.466 to 0.567] | 0.516 [0.450 to 0.592]
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-2: number analyzed (Participants) | 201 | 102
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-2 | 0.385 [0.359 to 0.414] | 0.467 [0.413 to 0.527]
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-3: number analyzed (Participants) | 201 | 102
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-3 | 0.426 [0.381 to 0.477] | 0.547 [0.472 to 0.633]
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-4: number analyzed (Participants) | 201 | 102
  Parent Trial Baseline Serostatus: Negative; Month 0 vs Parent Trial Month 9; DENV-4 | 0.557 [0.501 to 0.619] | 0.560 [0.494 to 0.634]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-1: number analyzed (Participants) | 154 | 43
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-1 | 0.403 [0.354 to 0.459] | 0.492 [0.378 to 0.641]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-2: number analyzed (Participants) | 154 | 43
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-2 | 0.259 [0.233 to 0.287] | 0.296 [0.242 to 0.362]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-3: number analyzed (Participants) | 154 | 43
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-3 | 0.387 [0.335 to 0.446] | 0.426 [0.327 to 0.556]
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-4: number analyzed (Participants) | 154 | 43
  Parent Trial Baseline Serostatus: Negative; Month 12 vs Parent Trial Month 9; DENV-4 | 0.359 [0.315 to 0.410] | 0.553 [0.416 to 0.734]

81. Secondary Outcome: GMR of Neutralizing Antibodies for Each of the 4 Dengue Serotypes in the Booster Phase
Description: The geometric mean ratio is the geometric mean of the ratio of the two visits being compared.
Time Frame: Months (M) 1&6 post-booster dose in current trial vs M 4 in parent trials; post-booster M 6 vs post-booster M 1; post-booster M 1 vs pre-booster (M 15 for DEN-304/M 42 for DEN-315); post-booster M 6 vs pre-booster (M 15 for DEN-304/M 42 for DEN-315)
Population: PPS-B included all participants from the FAS-B who received two doses of Takeda's TDV in the parent trials with no new major protocol violations after administration of the trial vaccination at Visit 3 that could potentially confound the primary endpoints in the current trial. Number analyzed: number of participants with data available for analysis for the specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
unitless ratio
  Booster Month 1 vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 95 | 94
  Booster Month 1 vs Parent Trial Month 4: DENV-1 | 0.352 [0.296 to 0.417] | 4.298 [3.204 to 5.767]
  Booster Month 1 vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 95 | 94
  Booster Month 1 vs Parent Trial Month 4: DENV-2 | 0.124 [0.107 to 0.144] | 0.378 [0.285 to 0.502]
  Booster Month 1 vs Parent Trial Month 4: DENV-3: number analyzed (Participants) | 95 | 94
  Booster Month 1 vs Parent Trial Month 4: DENV-3 | 0.231 [0.188 to 0.284] | 3.042 [2.217 to 4.175]
  Booster Month 1 vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 95 | 94
  Booster Month 1 vs Parent Trial Month 4: DENV-4 | 0.136 [0.107 to 0.174] | 1.505 [1.093 to 2.072]
  Booster Month 6 vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 92 | 89
  Booster Month 6 vs Parent Trial Month 4: DENV-1 | 0.285 [0.235 to 0.345] | 1.409 [1.036 to 1.917]
  Booster Month 6 vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 92 | 89
  Booster Month 6 vs Parent Trial Month 4: DENV-2 | 0.100 [0.086 to 0.117] | 0.206 [0.158 to 0.269]
  Booster Month 6 vs Parent Trial Month 4:DENV-3: number analyzed (Participants) | 92 | 89
  Booster Month 6 vs Parent Trial Month 4:DENV-3 | 0.225 [0.187 to 0.272] | 1.133 [0.816 to 1.573]
  Booster Month 6 vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 92 | 89
  Booster Month 6 vs Parent Trial Month 4: DENV-4 | 0.110 [0.088 to 0.137] | 0.468 [0.345 to 0.635]
  Booster Month 6 vs Booster Month 1: DENV-1: number analyzed (Participants) | 93 | 89
  Booster Month 6 vs Booster Month 1: DENV-1 | 0.817 [0.730 to 0.914] | 0.334 [0.283 to 0.395]
  Booster Month 6 vs Booster Month 1: DENV-2: number analyzed (Participants) | 93 | 89
  Booster Month 6 vs Booster Month 1: DENV-2 | 0.825 [0.753 to 0.903] | 0.535 [0.452 to 0.634]
  Booster Month 6 vs Booster Month 1: DENV-3: number analyzed (Participants) | 93 | 89
  Booster Month 6 vs Booster Month 1: DENV-3 | 0.990 [0.894 to 1.096] | 0.370 [0.295 to 0.463]
  Booster Month 6 vs Booster Month 1: DENV-4: number analyzed (Participants) | 93 | 89
  Booster Month 6 vs Booster Month 1: DENV-4 | 0.842 [0.744 to 0.954] | 0.323 [0.263 to 0.396]
  Booster Month 1 vs Pre-booster dose: DENV-1: number analyzed (Participants) | 99 | 97
  Booster Month 1 vs Pre-booster dose: DENV-1 | 0.962 [0.879 to 1.053] | 11.762 [8.660 to 15.975]
  Booster Month 1 vs Pre-booster dose: DENV-2: number analyzed (Participants) | 99 | 97
  Booster Month 1 vs Pre-booster dose: DENV-2 | 0.936 [0.862 to 1.016] | 2.822 [2.208 to 3.607]
  Booster Month 1 vs Pre-booster dose: DENV-3: number analyzed (Participants) | 99 | 97
  Booster Month 1 vs Pre-booster dose: DENV-3 | 0.856 [0.773 to 0.948] | 14.889 [10.992 to 20.170]
  Booster Month 1 vs Pre-booster dose: DENV-4: number analyzed (Participants) | 99 | 97
  Booster Month 1 vs Pre-booster dose: DENV-4 | 0.977 [0.855 to 1.117] | 13.162 [9.443 to 18.345]
  Booster Month 6 vs Pre-booster dose: DENV-1: number analyzed (Participants) | 96 | 92
  Booster Month 6 vs Pre-booster dose: DENV-1 | 0.784 [0.699 to 0.879] | 3.810 [2.847 to 5.097]
  Booster Month 6 vs Pre-booster dose: DENV-2: number analyzed (Participants) | 96 | 92
  Booster Month 6 vs Pre-booster dose: DENV-2 | 0.763 [0.697 to 0.835] | 1.550 [1.250 to 1.923]
  Booster Month 6 vs Pre-booster dose: DENV-3: number analyzed (Participants) | 96 | 92
  Booster Month 6 vs Pre-booster dose: DENV-3 | 0.858 [0.767 to 0.960] | 5.622 [4.151 to 7.614]
  Booster Month 6 vs Pre-booster dose: DENV-4: number analyzed (Participants) | 96 | 92
  Booster Month 6 vs Pre-booster dose: DENV-4 | 0.808 [0.703 to 0.929] | 4.289 [3.205 to 5.741]

82. Secondary Outcome: GMR of Neutralizing Antibodies for Each of the 4 Dengue Serotypes by Serostatus at Baseline in the Parent Trials in the Booster Phase
Description: as for outcome 80
Time Frame: Months (M) 1&6 post-booster dose in current trial vs M 4 in parent trials; post-booster M 1 vs pre-booster (M 15 for DEN-304/M 42 for DEN-315); post-booster M 6 vs pre-booster (M 15 for DEN-304/M 42 for DEN-315); post-booster M 6 vs post-booster M 1
Population: as for outcome 81
Measure: Geometric Mean (95% Confidence Interval); unit: unitless ratio
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 102 | 100
unitless ratio
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-1 | 0.413 [0.236 to 0.721] | 2.219 [1.181 to 4.169]
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-2 | 0.118 [0.077 to 0.180] | 0.355 [0.203 to 0.620]
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-3: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-3 | 0.311 [0.186 to 0.520] | 1.566 [0.684 to 3.583]
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Parent Trial Month 4: DENV-4 | 0.187 [0.111 to 0.315] | 1.018 [0.539 to 1.922]
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-1: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-1 | 1.033 [0.833 to 1.280] | 3.683 [1.612 to 8.412]
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-2: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-2 | 0.803 [0.615 to 1.049] | 1.805 [1.311 to 2.485]
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-3: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-3 | 0.825 [0.580 to 1.174] | 3.699 [1.738 to 7.873]
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-4: number analyzed (Participants) | 12 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 1 vs Pre-booster dose: DENV-4 | 1.310 [0.754 to 2.279] | 5.895 [2.657 to 13.078]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-1: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-1 | 1.065 [0.673 to 1.686] | 1.404 [0.787 to 2.506]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-2: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-2 | 0.739 [0.480 to 1.137] | 0.906 [0.673 to 1.221]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-3: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-3 | 0.965 [0.733 to 1.271] | 1.544 [0.868 to 2.748]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-4: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Pre-booster dose: DENV-4 | 0.871 [0.492 to 1.543] | 1.923 [0.941 to 3.931]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-1: number analyzed (Participants) | 9 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-1 | 0.998 [0.742 to 1.343] | 0.379 [0.221 to 0.650]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-2: number analyzed (Participants) | 9 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-2 | 1.026 [0.713 to 1.475] | 0.506 [0.330 to 0.775]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-3: number analyzed (Participants) | 9 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-3 | 1.024 [0.821 to 1.278] | 0.437 [0.255 to 0.750]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-4: number analyzed (Participants) | 9 | 11
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Booster Month 1: DENV-4 | 0.772 [0.462 to 1.292] | 0.349 [0.204 to 0.597]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4: DENV-1: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4: DENV-1 | 0.400 [0.175 to 0.915] | 0.779 [0.379 to 1.599]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4: DENV-2: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4: DENV-2 | 0.103 [0.066 to 0.162] | 0.161 [0.086 to 0.304]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4:DENV-3: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4:DENV-3 | 0.333 [0.215 to 0.515] | 0.593 [0.267 to 1.321]
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4: DENV-4: number analyzed (Participants) | 10 | 12
  Parent Trial Baseline Serostatus: Positive; Booster Month 6 vs Parent Trial Month 4: DENV-4 | 0.113 [0.063 to 0.201] | 0.314 [0.134 to 0.735]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-1: number analyzed (Participants) | 83 | 83
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-1 | 0.343 [0.286 to 0.413] | 4.692 [3.404 to 6.467]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-2: number analyzed (Participants) | 83 | 83
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-2 | 0.125 [0.106 to 0.147] | 0.382 [0.278 to 0.523]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-3: number analyzed (Participants) | 83 | 83
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-3 | 0.221 [0.177 to 0.277] | 3.322 [2.359 to 4.678]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-4: number analyzed (Participants) | 83 | 83
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Parent Trial Month 4; DENV-4 | 0.130 [0.099 to 0.171] | 1.585 [1.112 to 2.259]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-1: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-1 | 0.953 [0.862 to 1.053] | 13.646 [9.906 to 18.796]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-2: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-2 | 0.956 [0.876 to 1.043] | 2.988 [2.275 to 3.925]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-3: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-3 | 0.860 [0.771 to 0.959] | 17.792 [13.012 to 24.329]
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-4: number analyzed (Participants) | 87 | 86
  Parent Trial Baseline Serostatus: Negative; Booster Month 1 vs Pre-booster dose; DENV-4 | 0.939 [0.820 to 1.074] | 14.586 [10.186 to 20.888]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-1: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-1 | 0.756 [0.672 to 0.851] | 4.425 [3.233 to 6.056]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-2: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-2 | 0.766 [0.698 to 0.840] | 1.680 [1.321 to 2.137]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-3: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-3 | 0.846 [0.749 to 0.957] | 6.824 [4.957 to 9.395]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-4: number analyzed (Participants) | 86 | 80
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Pre-booster dose; DENV-4 | 0.801 [0.692 to 0.926] | 4.837 [3.533 to 6.623]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-1: number analyzed (Participants) | 84 | 78
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-1 | 0.799 [0.709 to 0.902] | 0.328 [0.274 to 0.393]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-2: number analyzed (Participants) | 84 | 78
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-2 | 0.805 [0.733 to 0.885] | 0.539 [0.447 to 0.650]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-3: number analyzed (Participants) | 84 | 78
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-3 | 0.986 [0.882 to 1.103] | 0.361 [0.282 to 0.463]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-4: number analyzed (Participants) | 84 | 78
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Booster Month 1; DENV-4 | 0.850 [0.746 to 0.969] | 0.319 [0.255 to 0.399]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-1: number analyzed (Participants) | 82 | 77
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-1 | 0.273 [0.224 to 0.333] | 1.546 [1.102 to 2.168]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-2: number analyzed (Participants) | 82 | 77
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-2 | 0.100 [0.085 to 0.118] | 0.214 [0.160 to 0.288]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-3: number analyzed (Participants) | 82 | 77
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-3 | 0.215 [0.175 to 0.263] | 1.253 [0.875 to 1.795]
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-4: number analyzed (Participants) | 82 | 77
  Parent Trial Baseline Serostatus: Negative; Booster Month 6 vs Parent Trial Month 4; DENV-4 | 0.109 [0.086 to 0.139] | 0.498 [0.357 to 0.694]

83. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) Within 7 Days Post-Booster Vaccination
Description: Solicited local AEs at injection site are defined as pain, erythema and swelling that occurred within 7 days post-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315). AEs were graded by the investigator in the following manner: Mild: Grade 1: Awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with everyday activities. Relieved with or without symptomatic treatment; Moderate: Grade 2: Sufficient discomfort is present to cause interference with normal activity. Only partially relieved with symptomatic treatment; Severe: Grade 3: Extreme distress, causing significant impairment of functioning or incapacitation. Prevents normal everyday activities. Not relieved with symptomatic treatment.
Time Frame: Days 1 through 7 post-booster dose at Visit 3 (Month 15 [DEN-304]) and (Month 42 [DEN-315])
Population: Safety Set-Booster (SAF-B) included all participants who received at least one dose of Takeda's TDV in the parent trials and who received the trial vaccination in the current trial. Overall number of participants analyzed: number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 115 | 112
percentage of participants
  Mild | 17.4 | 50.0
  Moderate | 5.2 | 14.3
  Severe | 0 | 1.8

84. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events Within 14 Days Post-Booster Vaccination by Severity
Description: Solicited systemic AEs are defined as fever, headache, asthenia, malaise and myalgia that occurred within 14 days post-booster dose at Month 15 (DEN-304) and Month 42 (DEN-315). AEs were graded by the investigator in the following manner: Mild: Grade 1: Awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with everyday activities. Relieved with or without symptomatic treatment; Moderate: Grade 2: Sufficient discomfort is present to cause interference with normal activity. Only partially relieved with symptomatic treatment; Severe: Grade 3: Extreme distress, causing significant impairment of functioning or incapacitation. Prevents normal everyday activities. Not relieved with symptomatic treatment.
Time Frame: Days 1 through 14 post-booster dose at Visit 3 (Month 15 [DEN-304]) and (Month 42 [DEN-315])
Population: SAF-B included all participants who received at least one dose of Takeda's TDV in the parent trials and who received the trial vaccination in the current trial. Overall number of participants analyzed: number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 115 | 112
percentage of participants
  Mild | 30.4 | 32.1
  Moderate | 12.2 | 17.0
  Severe | 1.7 | 3.6

85. Secondary Outcome: Percentage of Participants With Any Unsolicited AEs in the Booster Phase
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine or placebo; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Days 1 through 28 post-booster dose at Visit 3 (Month 15 [DEN-304]) and (Month 42 [DEN-315])
Population: SAF-B included all participants who received at least one dose of Takeda's TDV in the parent trials and who received the trial vaccination in the current trial.
Measure: Number; unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 118 | 115
percentage of participants | 6.8 | 6.1

86. Secondary Outcome: Percentage of Participants With Any Medically Attended AEs (MAAEs) in the Booster Phase
Description: MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: Month 15 post-booster dose through Month 21 (DEN-304); Month 42 post-booster dose through Month 48 (DEN-315)
Population: as for outcome 85
Measure: Number; unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 118 | 115
percentage of participants | 16.9 | 11.3

87. Secondary Outcome: Percentage of Participants With Any Serious Adverse Events (SAEs) Prior to the Booster Dose
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine or placebo; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined as any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically important event.
Time Frame: Month 0 through Month 15 (DEN-304) and Month 42 (DEN-315)
Population: SAF included all participants who agreed to participate in the current trial, did not screen fail, and who received at least one dose of Takeda's TDV in the parent trials.
Measure: Number; unit: percentage of participants
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315
Number analyzed (Participants) | 246 | 119
percentage of participants | 2.4 | 6.7

88. Secondary Outcome: Percentage of Participants With Any SAEs in the Booster Phase
Description: as for outcome 87
Time Frame: Month 15 post-booster dose after vaccination through Month 21 (DEN-304); Month 42 post-booster dose after vaccination through Month 48 (DEN-315)
Population: as for outcome 85
Measure: Number; unit: percentage of participants
Arm/Group | Booster Phase: Placebo | Booster Phase: TDV
Number analyzed (Participants) | 118 | 115
percentage of participants | 2.5 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality & SAEs: From Day 1 [Month 0] up to Month 21 (DEN-304) & Month 48 (DEN-315); Non-serious adverse events: Up to 28 days (day of vaccination + 27 days) after administration of each vaccine dose on Months 15 (DEN-304) & 42 (DEN-315).
Description: Prior to Booster Arms: SAF included all participants who agreed to participate in current trial,did not screen fail& who received at least 1 dose of Takeda's TDV in parent trials.
  Booster Phase Arms: SAF-B included all participants who received at least 1 dose of Takeda's TDV in parent trials &who received the trial vaccination in current trial.
Groups:
- Booster Phase: TDV: Participants received TDV 0.5 mL, injection, subcutaneously, once at Month 15 for participants from parent trials DEN-304 (US) or once at Month 42 for participants from parent trial DEN-315 (Mexico).
- Booster Phase: Placebo: Participants received TDV placebo-matching 0.5 mL injection, subcutaneously, once at Month 15 for participants from parent trial DEN-304 (US) or once at Month 42 for participants from parent trial DEN-315 (Mexico).
Arm/Group | Prior to Booster: DEN-304 | Prior to Booster: DEN-315 | Booster Phase: TDV | Booster Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/246 | 1/119 | 0/115 | 0/118
Serious Adverse Events (participants affected / at risk) | 6/246 | 8/119 | 0/115 | 3/118
Other Adverse Events (participants affected / at risk) | 0/246 | 0/119 | 83/115 | 57/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior to Booster: DEN-304 (N=246) | Prior to Booster: DEN-315 (N=119) | Booster Phase: TDV (N=115) | Booster Phase: Placebo (N=118)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pilonidal disease (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior to Booster: DEN-304 (N=246) | Prior to Booster: DEN-315 (N=119) | Booster Phase: TDV (N=115) | Booster Phase: Placebo (N=118)
Asthenia (General disorders) | 0 | 0 | 28 | 22
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 29 | 0
Headache (Nervous system disorders) | 0 | 0 | 42 | 38
Injection site erythema (General disorders) | 0 | 0 | 8 | 2
Malaise (General disorders) | 0 | 0 | 28 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 40 | 22
Pain (General disorders) | 0 | 0 | 70 | 26
Swelling (General disorders) | 0 | 0 | 16 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03999996/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT03999996/SAP_001.pdf